CLINICAL TRIAL: NCT01335126
Title: Comparison of Tolerability and Clinical Performance of Two Emulsion-type Artificial Tears
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hom, Milton M., OD, FAAO (Individual)
Collaborators: Allergan (Industry)
Responsible Party: Milton M. Hom, OD, FAAO., Private Practice
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AG9965-007
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Dry Eye
Keywords: Artificial tears
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Test (Experimental)
  Interventions: Other: Emulsion type artificial tear

INTERVENTIONS:
Other: Emulsion type artificial tear — 2 types of artificial tears

SUMMARY:
The purpose of this study is to evaluate the performance between two emulsion-type artificial tears.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and over inclusive.
* Males or females
* Patient is in generally good & stable overall health.
* Patient likely to comply with study guidelines & study visits.
* Informed consent signed.
* OSDI score >18 OR
* TBUT <10 seconds

Exclusion Criteria:

* Corneal refractive surgery or contact lens wear within 6 months of this study.
* Current use of Restasis
* Intra-ocular surgery within 6 months or ocular laser surgery within 6 months.
* Pregnant or lactating women.
* Ocular pathology (includes glaucoma and cataract), which could impact results and/or place patient at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-10 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Tolerability Questionnaire | 8 weeks
  Tolerability (comfort) measured with Visual Analog scale (1 to 100)

SECONDARY OUTCOMES:
Acceptability Questionnaire | 8 weeks
  Acceptability questionnaire on statements regarding drop satisfaction, etc. Answered as A to E (Strongly Agree, Agree, Neither Agree or Disagree, Disagree or Strongly Disagree)
Tear Break Up Time | 2-3 weeks
  Tear Break Up Time measured in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Milton M Hom, OD FAAO, Principal Investigator — Private Practice